CLINICAL TRIAL: NCT01324973
Title: Web-Based Weight Management for Individuals With Mental Illness
Acronym: eWellness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Los Angeles County Department of Mental Health (Unknown); University of Maryland (Other)
Responsible Party: Principal Investigator, Alexander S. Young, MD MSHS, Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5R34MH090207 (NIH)
Record Dates: First submitted 2011-03-28; First posted 2011-03-29 (Estimated); Last update posted 2014-07-02 (Estimated); Status verified 2014-06

CONDITIONS: Mental Disorders; Schizophrenia; Affective Disorders, Psychotic; Overweight; Obesity
Keywords: Medical Informatics; Therapy, Computer-Assisted; Health Education; Diet; Exercise
MeSH Terms: conditions — Mental Disorders; Schizophrenia; Affective Disorders, Psychotic; Overweight; Obesity; Health Education; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- eWellness program (Experimental): A comprehensive program that delivers web-based, evidence-based weight management; and structured peer supports. The program is designed to meet the needs of individuals with mental illness.
  Interventions: Behavioral: eWellness
- Control group (No Intervention): Care as usual

INTERVENTIONS:
Behavioral: eWellness — A weight management program that includes computerized delivery of evidence-based education regarding diet and physical activity, and peer coaching.
  Other Names: web-based weight management with peer coaching
  Arms: eWellness program

SUMMARY:
Obesity and physical inactivity have become serious problems for individuals with mental illness, resulting in increased rates of chronic disease, premature death, and substantial health care costs. Although in-person psychoeducational interventions help individuals with mental illness manage their weight, these interventions are often not used because they require frequent travel to treatment programs and substantial time from clinicians. This project addresses these barriers by developing and evaluating the effectiveness of an web-based computer system that is focused on diet and exercise education, and designed to help individuals with mental illness manage their weight.

DETAILED DESCRIPTION:
Background/Rationale: Obesity and physical inactivity have reached epidemic proportions, resulting in increased rates of chronic disease, premature death, and substantial health care costs. Excess weight is even more prevalent in populations with serious mental illnesses (SMI), in part due to medication-induced weight gain and social disadvantage. Since individuals with SMI often have cognitive deficits, specialized approaches are required to help people manage their weight. Researchers have found that specialized in-person interventions focused on diet and activity can help individuals with SMI manage their weight. However, these evidence-based practices have not been widely disseminated. Barriers to the use of these interventions include reluctance of individuals to participate in groups, difficulty finding transportation for frequent visits to clinics, a shortage of trained clinicians, and inadequate clinician time to provide the interventions. It is likely that these barriers can be addressed with a web-based weight intervention that is tailored for individuals with SMI. Specialized web-based approaches have been studied and found to be effective in this population, and can deliver content that is intensive and engaging with minimal requirements for clinician time.

Objectives: The investigators on this proposal previously developed a prototype web-based system that provides limited diet education to individuals with SMI. The current project extends and evaluates this system. The project's objectives are to: 1) build on the prototype to develop "eWellness," a comprehensive web-based system that delivers an evidence-based weight management program focused on diet and activity, and that meets the needs of individuals with SMI; 2) evaluate the effectiveness, in individuals with SMI, of an eWellness program compared with a control group; and, 3) characterize, from the perspective of individuals with SMI, the strengths, weaknesses, and barriers to the use of eWellness.

Methods: This is a randomized, controlled trial of individuals with SMI at a community mental health center who are overweight and prescribed medications that have weight gain as a common side-effect. Participants are assigned to the eWellness program or to continue with usual care. Research assessments occur at baseline, 3, and 6 months. Changes in outcomes are compared over time between the two groups.

Significance: By losing weight, individuals with mental illness can decrease their risk for medical problems, and improve their quality of life and life expectancy. A web-based system that helps individuals lose weight could be feasible to disseminate broadly at medical centers, clinics, and community based programs in both rural and urban areas.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of schizophrenia, schizoaffective disorder, bipolar disorder, recurrent major depressive disorder with psychosis, or chronic PTSD
* age 18 and over
* prescribed antipsychotic medication for at least 3 months
* BMI of 30 or higher, or BMI of 28 or higher if 10 pounds of recent weight gain
* medical clearance to participate
* control over diet

Exclusion Criteria:

* any medical condition for which a weight program is contraindicated
* history of bariatric surgery
* psychiatric hospitalization during the prior month
* pregnant and nursing mothers
* diagnosis of dementia
* not able to provide informed consent by self or legally appointed representative

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-03; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
dietary habits | 6 months
physical activity | 6 months
weight | 6 months
waist circumference | 6 months
diet and activity-related self-efficacy, motivation, and readiness to change | 6 months

SECONDARY OUTCOMES:
health-related functioning | 6 months
quality of life | 6 months
strengths, weaknesses, and barriers to the use of eWellness | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Alexander S Young, MD, MSHS, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Center for Health Services and Society, Los Angeles, California, United States

REFERENCES:
- [Background] Chinman M, Young AS, Schell T, Hassell J, Mintz J. Computer-assisted self-assessment in persons with severe mental illness. J Clin Psychiatry. 2004 Oct;65(10):1343-51. doi: 10.4088/jcp.v65n1008. PMID 15491237
- [Background] Chinman M, Hassell J, Magnabosco J, Nowlin-Finch N, Marusak S, Young AS. The feasibility of computerized patient self-assessment at mental health clinics. Adm Policy Ment Health. 2007 Jul;34(4):401-9. doi: 10.1007/s10488-007-0120-4. Epub 2007 Apr 24. PMID 17453332
- [Background] Young AS, Chaney E, Shoai R, Bonner L, Cohen AN, Doebbeling B, Dorr D, Goldstein MK, Kerr E, Nichol P, Perrin R. Information technology to support improved care for chronic illness. J Gen Intern Med. 2007 Dec;22 Suppl 3(Suppl 3):425-30. doi: 10.1007/s11606-007-0303-4. PMID 18026812
- [Background] Young AS. The client, the clinician, and the computer. Psychiatr Serv. 2010 Jul;61(7):643. doi: 10.1176/ps.2010.61.7.643. No abstract available. PMID 20591993
- [Background] Cohen AN, Chinman MJ, Hamilton AB, Whelan F, Young AS. Using patient-facing kiosks to support quality improvement at mental health clinics. Med Care. 2013 Mar;51(3 Suppl 1):S13-20. doi: 10.1097/MLR.0b013e31827da859. PMID 23407006
- [Background] Hamilton AB, Chinman M, Cohen AN, Oberman RS, Young AS. Implementation of consumer providers into mental health intensive case management teams. J Behav Health Serv Res. 2015 Jan;42(1):100-8. doi: 10.1007/s11414-013-9365-8. PMID 24091610
- [Background] Niv N, Cohen AN, Hamilton A, Reist C, Young AS. Effectiveness of a psychosocial weight management program for individuals with schizophrenia. J Behav Health Serv Res. 2014 Jul;41(3):370-80. doi: 10.1007/s11414-012-9273-3. PMID 22430566
- [Result] Cohen AN, Golden JF, Young AS. Peer wellness coaches for adults with mental illness. Psychiatr Serv. 2014 Jan 1;65(1):129-30. doi: 10.1176/appi.ps.650101. No abstract available. PMID 24382767